CLINICAL TRIAL: NCT00561496
Title: Single Dose and 14-Day Once or Twice-Daily Pharmacokinetic Study of the Vaginal Microbicide Agent 1% Tenofovir Gel
Brief Title: Pharmacokinetic Study of the Vaginal Microbicide Agent 1% Tenofovir Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Collaborators: International Partnership for Microbicides, Inc. (Industry); Gilead Sciences (Industry)
Responsible Party: Jill Schwartz, MD/Project Leader, CONRAD
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A04-095
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections
Keywords: HIV prevention; Microbicides; Pharmacokinetics; vaginal biopsies
MeSH Terms: conditions — HIV Infections | interventions — Adenine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Twice daily (Other): Tenofovir gel intravaginal twice daily for 14 days
  Interventions: Drug: Tenofovir gel
- Once daily (Other): Tenofovir gel intravaginal once daily for 14 days
  Interventions: Drug: Tenofovir gel

INTERVENTIONS:
Drug: Tenofovir gel — Intravaginal (4grams)single dose followed by fourteen days
  Other Names: 9-[(R)-2-(phosphonomethoxy)propyl] adenine or PMPA

SUMMARY:
This is a multi-center, pharmacokinetic study involving a single-dose phase, a wash out phase and a two-week once or twice-daily dosing phase for each of 49 volunteers.

In the single-dose phase, each volunteer will apply the single dose in the clinic. Participants will be randomized to have cervicovaginal samples and biopsies collected at one of seven time-points [0.5, 1, 2, 4, 6, 8, and 24 hour(s)] after the single-dose. Blood samples will be drawn at 0.5, 1, 2, 4, 6, 8, and 24 hour(s) after the single-dose.

In the two-week phase, the study supplies will be distributed and the participants will be randomized to apply each dose either once or twice-daily for two weeks. At the one week follow-up visit a blood sample will be drawn prior to the morning dose to obtain a trough value and cervicovaginal samples will be collected four hours after the morning dose. At the two week follow-up visit blood samples will be drawn prior to the morning dose to obtain a trough value and then at 0.5, 1, 2, 4, 6, 8, and 24 hour(s) from the final morning dose. Participants will be randomized to have cervicovaginal samples and biopsies collected at either 4, 8 or 24 hours after the final morning dose.

Up to 10 participants who have completed the first two phases of the study, will be asked to participate in a third phase to have cervicovaginal samples, biopsies and blood samples collected 12 hours after a single-dose.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 18-45 years old, inclusive
* Must be in general good health by volunteer history without any clinically significant systemic disease (including liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease)
* Must have regular menstrual cycles (minimum of 26 and maximum of 38 days)
* Must be at least 2 months since last pregnancy outcome and have had at least two spontaneous menses
* Must abstain from sexual activity and use of intravaginal products for 72 hours prior to the start of the single-dose phase and multi-dose phase, for at least one week following vaginal biopsies and for the duration of the study phases
* Willingness to give voluntary consent, sign an informed consent form and comply with study procedures as required by the protocol

Exclusion Criteria:

* Currently pregnant or at risk for pregnancy (may be using Paragard® IUD, effective barrier method, female sterilization or abstinence, or be sexually active with a vasectomized partner)
* Currently breastfeeding or planning to breastfeed during the course of the study
* Use of any hormonal contraceptives within 30 days of enrollment
* Use of Depo-Provera within 120 days of enrollment History of abnormal Pap smear (by volunteer history) that has not been evaluated and treated, if indicated, according to standard guidelines
* Current vaginal or urinary tract infection
* Positive test for Neisseria gonorrhea or Chlamydia trachomatis at the time of screening
* Positive wet mount for Trichomonas vaginalis at the time of screening or enrollment
* Deep epithelial genital findings such as abrasions, ulcerations, and lacerations, or vesicles suspicious for a sexually transmitted infection
* Current or past use of any anti-retroviral therapies including but not limited to systemic tenofovir (Viread®)
* Current or recent drug or alcohol abuse
* Current or anticipated use of drugs on a daily basis that may reduce renal function (e.g. acyclovir or ibuprofen) or liver function (e.g. tylenol)
* HIV positive at the time of screening
* Hepatitis B surface antigen (HBsAg) positive at the time of screening
* Grade 1 or higher serum chemistry or complete blood count abnormality in accordance with DAIDS toxicity table values
* Abnormal finding on laboratory or physical examination or a medical condition which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data
* Participation in any other research study in the 30 days prior to screening and/or plans to participate in any other research study during entire study duration

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Concentration of tenofovir in local genital tract compartments (intraluminal, mononuclear cells and vaginal tissue levels). Concentration (Cmax) and time of maximum concentration (Tmax) of tenofovir in the systemic compartment. | Single dose; two weeks (after once or twice-daily vaginal administration)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Schwartz, MD, Study Director — CONRAD
Locations (3):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Advances in Health, Inc, Houston, Texas
- Profamilia, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Schwartz JL, Rountree W, Kashuba AD, Brache V, Creinin MD, Poindexter A, Kearney BP. A multi-compartment, single and multiple dose pharmacokinetic study of the vaginal candidate microbicide 1% tenofovir gel. PLoS One. 2011;6(10):e25974. doi: 10.1371/journal.pone.0025974. Epub 2011 Oct 19. PMID 22039430